CLINICAL TRIAL: NCT05593016
Title: Improving Symptom Management for Adolescents and Young Adults With Advanced Cancer: Development and Pilot Testing of a Novel Intervention
Brief Title: Adolescents and Young Adults (AYAs) With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110574; R21CA263727-01A1 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-10-25 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Adolescent and Young Adult Cancer Patient
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) (Experimental): Four, 60-minute sessions will provide training on behavioral symptom management skills, delivered over 6-8 weeks to patients in their homes using videoconferencing.
  Interventions: Behavioral: Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
- Education Control Arm (Experimental): The control arm will receive the NCI booklet, "Taking Time: Support for People with Cancer" and otherwise continue their usual care.
  Interventions: Behavioral: Education Control Arm

INTERVENTIONS:
Behavioral: Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) — Participating in the SMILE arm of the study will consist of four, 60-minute sessions delivered over 6-8 weeks to patients in their homes using videoconferencing.
  Intervention will provide training in behavioral symptom management skills (e.g.,relaxation training, activity-rest cycling) and include skills from ACT and MCP targeting avoidance of uncomfortable experiences (e.g., thoughts, emotions) and promoting engagement in value-directed activity.
  Arms: Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
Behavioral: Education Control Arm — The control arm will receive the NCI booklet, "Taking Time: Support for People with Cancer," which provides basic strategies for symptom (e.g., pain, fatigue, stress) management, coping with negative emotions, and communication and will continue their usual medical care of advanced cancer.
  Arms: Education Control Arm

SUMMARY:
This study aims to develop and test the feasibility and acceptability of a psychosocial symptom management intervention designed to meet the unique needs of Adolescents and Young Adults (AYAs) with advanced cancer. The proposed intervention will combine traditional behavioral symptom management strategies commonly use in the palliative care setting with important skills and concepts from Meaning-Centered Psychotherapy and Acceptance and Commitment Therapy. Skills from these approaches may be particularly relevant to AYAs with advanced cancer who experience significant disruption in life goals from cancer and associated symptoms and may have greater difficulties understanding and finding meaning in their lives than older and younger patients. Intervention content, structure, and study procedures will be informed by qualitative data obtained during interviews/focus groups with patient (n=16) and caregiver (n=12) stakeholders as well as review by patient user testers (n=3). It is anticipated that the intervention will include four weekly sessions spaced over 6-8 weeks and be delivered using videoconferencing. Next, AYAs with advanced cancer (N=40) will be randomized to the intervention or education control arms using an allocation ratio of 1.5: 1. The study team will examine the feasibility of study recruitment and retention, acceptability, and changes in variables of interest (i.e., physical and psychological symptoms, symptom interference, self-efficacy for symptom management, experiential avoidance, values) over time for the intervention and control arms. Participants will also provide feedback on study materials, intervention format, and the appropriateness of the intervention to the population and advanced stage of disease.

DETAILED DESCRIPTION:
The investigators propose to begin to fill this gap by developing and pilot testing a psychosocial symptom management intervention designed to meet the unique needs of AYAs with advanced cancer. Guided by the team's prior work developing symptom management interventions for older advanced cancer patients and expertise in AYA Oncology, the proposed intervention will combine traditional behavioral symptom management strategies (e.g., activity pacing, relaxation training) commonly used in palliative care with important skills and concepts from Meaning-Centered Psychotherapy (MCP) and Acceptance and Commitment Therapy (ACT). Both MCP and ACT have been associated with decreased distress and symptom burden in oncology patients with advanced cancer. The study team anticipates that the intervention will incorporate questions from MCP to help patients identify valued life areas impacted by symptoms; techniques from ACT will then be used to help patients obtain distance from psychological barriers (e.g., thoughts, emotional experiences) to enacting their values to allow for flexible, value-congruent behaviors. Skills from these approaches may be particularly relevant to AYAs with advanced cancer who experience significant disruption in life goals due to symptoms and may have greater difficulty understanding and finding meaning in their lives.

Aim 1: Intervention Development. Preliminary intervention content has been outlined and will be further informed by interviews with patients (AYAs with advanced cancer, aged 15-29; two groups, n=12), caregivers (one group, n=8), and a combined patient/caregiver group (one group; AYAs: n=4; caregivers: n=4) who will provide information about the symptom (e.g., pain, fatigue, emotional distress) experience of AYAs with advanced cancer, patients' symptom management needs and coping strategies, the unique developmental aspects of being an AYA or caring for an AYA with advanced cancer, and how patient and caregiver needs may interact to impact symptom management. Participant input will help to confirm whether the proposed intervention strategies (i.e., behavioral symptom management, ACT, MCP) may be of benefit for addressing the unique needs of AYAs with advanced cancer. User testing of the developed intervention will be conducted with an additional three AYAs with advanced cancer to further refine the intervention content and format, written study materials, and study procedures.

Aim 2: Pilot Randomized Controlled Trial. AYAs with advanced cancer (N=40) will be randomized to the intervention or an education control arm using an allocation ratio of 1.5:1. Feasibility of study recruitment (N=40 in 12 months) and participant retention (>80% intervention completion) will be examined along with intervention acceptability. Patterns of change in symptom (i.e., pain, fatigue, distress) severity and interference, self-efficacy for symptom management, and targets of ACT and MCP (e.g., acceptance, experiential avoidance, congruency between values and actions) will be examined.

This pilot trial will allow the study team to refine approaches to identify, recruit, and retain AYA participants and examine patterns of change in key outcome variables for the intervention and control arms. Information obtained will position the investigative team to examine the efficacy of the intervention in a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 15-29 years old
* Diagnosis of advanced (i.e., diagnosis of incurable cancer or distant metastases) or recurrent cancer
* Able to speak/read English

Exclusion Criteria:

* Active serious mental illness (e.g., schizophrenia)
* Visual, hearing, or cognitive impairment

Focus Group Caregiver Inclusion Criteria:

* 18 years old and older
* Ability to speak/read English

Focus Group Caregiver Exclusion Criteria:

* Visual, hearing or cognitive impairment
* Severe mental illness

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Dorfman, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two consented participants were lost to follow-up prior to completing the baseline assessment and were not randomized.
Groups:
- Intervention Development (Patients): Participants in this early stage of the study helped us to develop and refine the program that we subsequently used for the randomized controlled trial. These participants were patients who provided feedback on the program.
- Intervention Development (Caregivers): Participants in this early stage of the study helped us to develop and refine the program that we subsequently used for the randomized controlled trial. These participants were caregivers who provided feedback on the program.
- Intervention Refinement: Participants in this early stage of the study helped us to develop and refine the program that we subsequently used for the randomized controlled trial. These participants were patients who tested the first iteration of the program and provided feedback.
Period: Overall Study
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm | Intervention Development (Patients) | Intervention Development (Caregivers) | Intervention Refinement
Started | 24 | 16 | 17 | 13 | 3
Intervention Development | 0 | 0 | 17 | 13 | 0
Intervention Refinement | 0 | 0 | 0 | 0 | 3
Intervention Implementation | 24 | 16 | 0 | 0 | 0
Completed | 22 | 14 | 15 | 11 | 3
Not Completed | 2 | 2 | 2 | 2 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm | Intervention Development (Patients) | Intervention Development (Caregivers) | Intervention Refinement | Total
Number analyzed (Participants) | 24 | 16 | 17 | 13 | 3 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.42 (3.68) | 23.56 (3.93) | 23.47 (4.03) | 49.38 (11.41) | 23.00 (4.36) | 28.21 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 4 | 10 | 3 | 41
  Male | 8 | 8 | 13 | 3 | 0 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 13 | 1 | 0 | 0 | 17
  Not Hispanic or Latino | 21 | 2 | 16 | 12 | 3 | 54
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 4 | 4 | 4 | 2 | 0 | 14
  White | 16 | 11 | 13 | 9 | 3 | 52
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Acceptability Questionnaire
Description: The Treatment Acceptability Questionnaire is a six-item scale assessing participants' views of an intervention as acceptable, ethical, and effective. Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable") and averaged.
Time Frame: Post-treatment (6-8 weeks following the baseline assessment)
Population: This measure was only provided to participants who received the SMILE Intervention and analyzed among participants receiving at least one AYA SMILE session (n=20) were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
Number analyzed (Participants) | 20
score on a scale | 6.02 (0.76)

2. Primary Outcome: Session Attendance Percentage
Description: Treatment feasibility will be assessed by measuring the session attendance percentage for each participant receiving the intervention.
Time Frame: Post-treatment (6-8 weeks following the baseline assessment)
Population: Outcome only applicable to the SMILE Intervention arm.
Measure: Mean (Standard Deviation); unit: percentage of sessions
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
Number analyzed (Participants) | 24
percentage of sessions | 80.20 (39.69)

3. Primary Outcome: Study Enrollment (Randomized Controlled Trial)
Description: Number of participants who enrolled in the randomized controlled trial phase of the study after being found eligible.
Time Frame: 12 months following the start of study enrollment
Population: This measure is for individuals who were eligible for the randomized controlled trial. Only patients who were screened for eligibility to participate in the randomized controlled trial are included in this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Individuals who were eligible for the study.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 97
Participants | 42

4. Primary Outcome: Pain Severity as Measured by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory is a 9-item, self-report measure assessing pain severity and interference from pain across important life domains (e.g., general activity, work, relations with others). Participants rate their pain on a scale from 0 "no pain" to 10 "pain as bad as you can imagine." Pain severity is calculated as the average of four items assessing participants' worst, least, current, and average (in the last week) pain on a scale from 0 "no pain" to 10 "worst pain."
Time Frame: Baseline, post-treatment/follow-up (6-8 weeks following the baseline assessment), 4 weeks following the post-treatment/follow-up assessment; baseline and post-treatment (6-8 weeks following the baseline assessment) reported
Population: SMILE Intervention: One participant lost to follow-up, one participant with missing data; Education Control Arm: One participant lost to follow-up, one participant with missing data, and one participant died prior to completion of the A2 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 22 | 13
score on a scale
  Baseline | 2.49 (2.35) | 2.10 (1.89)
  Post-treatment | 2.28 (1.85) | 2.25 (1.88)

5. Primary Outcome: Pain Interference as Measured by the Brief Pain Inventory (BPI)
Description: The Brief Pain Inventory is a 9-item, self-report measure assessing pain severity and interference from pain across important life domains (e.g., general activity, work, relations with others). Pain interference is computed as the average of seven items, which ask about the interference of pain across different life domains (e.g., general activity, mood, relations with other people) in the past week on a scale from 0 "Does not interfere" to 10 "Completely interferes." Higher scores indicate higher levels of pain interference.
Time Frame: as for outcome 4
Population: SMILE Intervention: One participant lost to follow-up; Education Control Arm: One participant lost to follow-up and one participant died prior to completion of the A2 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
score on a scale
  Baseline | 2.53 (2.30) | 2.45 (2.66)
  Post-treatment | 1.91 (2.04) | 2.07 (2.60)

6. Primary Outcome: Fatigue as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: Fatigue will be assessed using the PROMIS Computer Adaptive Test for Fatigue. Questions ask participants to rate their fatigue during the past 7 days. The T-score ranges from 0 to 100, where higher T-scores indicate greater fatigue. Scores are converted to standardized t-scores with a mean of 50 and standard deviation of 10. T-scores of 55 to <60 indicate mild levels of fatigue, ≥60 to <70 indicates moderate levels of fatigue, and ≥70 indicate severe levels of fatigue.
Time Frame: as for outcome 4
Population: SMILE Intervention: One participant lost to follow-up; Education Control Arm: One participant lost to follow-up one participant died prior to completion of the A2 assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
T-score
  Baseline | 58.64 (9.39) | 54.23 (8.87)
  Post-treatment | 54.67 (8.12) | 51.24 (8.99)

7. Primary Outcome: Depressive Symptoms as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: Depressive Symptoms will be assessed using the PROMIS Computer Adaptive Test for Depression. Questions ask participants to respond to questions during the past 7 days. Scores are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher T-scores indicate higher levels of depression. T-scores of 55 to <60 indicate mild levels of depression, ≥60 to <70 indicates moderate levels of depression, and ≥70 indicate severe levels of depression.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
T-score
  Baseline | 56.15 (7.56) | 52.95 (10.28)
  Post-treatment | 51.35 (8.73) | 52.06 (10.41)

8. Primary Outcome: Self-Efficacy as Measured by the Managing Chronic Disease Scale
Description: The Self-Efficacy for Managing Chronic Disease Scale is a 6-item scale. Participants rate their confidence in keeping pain, fatigue, emotional distress, and other symptoms from interfering with things they want to do on a scale from 1 "not at all confident" to 10 "totally confident." The score for the scale is the mean of the six items, with higher number indicating higher self-efficacy.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
score on a scale
  Baseline | 6.75 (1.88) | 7.00 (2.19)
  Post-treatment | 7.89 (1.65) | 6.90 (2.17)

9. Primary Outcome: Acceptance and Action
Description: 7-Item: The Acceptance and Action Questionnaire-II assesses acceptance, experiential avoidance and psychological flexibility. Question scale ranges from 1, never true, to 7, always true. The total score ranges from 7 to 49, where a higher score indicates greater psychological inflexibility.
Time Frame: as for outcome 4
Population: SMILE Intervention: One participant lost to follow-up and two participants with missing data on at least one item of the subscale; Education Control Arm: One participant lost to follow-up and one participant died prior to completion of the A2 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 21 | 14
score on a scale
  Baseline | 21.19 (10.25) | 17.50 (9.15)
  Post-treatment | 19.19 (9.91) | 18.43 (8.25)

10. Primary Outcome: Spritual Well-Being: Functional Assessment of Chronic Illness Therapy (FACIT)
Description: The FACIT assesses the spiritual wellbeing of participants with 12-item questionnaire. Responses for each item are on a scale from 0 = "not at all" to 4 = "very much." Three subscale scores (Meaning, Peace, Faith) are calculated by summing specific items. Each subscale has 4 items, with total scores ranging from 0 to 16, with higher scores indicating greater well-being for each subscale (Meaning, Peace, or Faith). A total score is calculated as the sum of the three subscores, with total scores ranging from 0 to 48. Higher scores represent greater spiritual wellbeing.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
score on a scale
  Baseline: Meaning | 11.61 (3.93) | 12.5 (3.03)
  Post-treatment: Meaning | 12.48 (2.53) | 11.0 (4.54)
  Baseline: Peace | 8.87 (3.77) | 9.29 (4.08)
  Post-treatment: Peace | 10.28 (3.73) | 8.50 (4.47)
  Baseline: Faith | 9.87 (5.81) | 8.43 (5.33)
  Post-treatment: Faith | 11.35 (5.07) | 8.50 (4.96)
  Baseline: Total | 30.35 (10.51) | 30.21 (10.22)
  Post-treatment: Total | 34.10 (10.39) | 28.00 (12.31)

11. Primary Outcome: Anxiety Symptoms as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The PROMIS Computer Adaptive Test for Anxiety will be used to assess anxiety symptoms in the last week. Scores are converted to standardized T-scores with a mean of 50 and standard deviation of 10. Higher T-scores indicate higher levels of anxiety. T-scores of 55 to <60 indicate mild levels of anxiety, ≥60 to <70 indicates moderate levels of anxiety, and ≥70 indicate severe levels of anxiety.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 23 | 14
T-score
  Baseline | 58.06 (10.44) | 56.64 (10.48)
  Post-treatment | 53.81 (9.73) | 53.91 (10.40)

12. Primary Outcome: Intervention Satisfaction as Measured by the Satisfaction With Therapy and Therapist-Revised (SSTS-R)
Description: The SSTS-R is a 13-item measure. The first 12-items ask participants to rate their satisfaction with the therapy received (6-items) or the therapist delivering the intervention (6-items) on a five-point scale ranging from 1 "strongly disagree" to 5 "strongly disagree." Each of the subscales (Satisfaction With Therapy and Satisfaction With Therapist) range from 6 to 30, with higher scores indicating greater satisfaction. The 13th item (Global Improvement) asks, "How much did the intervention help with your symptoms?" with 5 answer choices ranging from 1 "made things a lot worse" to 5 "made things a lot better," where higher scores indicate a better outcome.
Time Frame: Post-treatment (6-8 weeks following the baseline assessment)
Population: Only participants receiving one intervention session had data analyzed. One of these participants had missing data on this item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
Number analyzed (Participants) | 19
score on a scale
  Satisfaction with therapy subscale | 26.42 (2.81)
  Satisfaction with therapist subscale | 27.57 (3.10)
  How much did this intervention help with symptoms? | 4.40 (0.50)

13. Primary Outcome: Values as Measured by the Bulls Eye Values Survey
Description: The Bulls Eye Values Survey assists participants with clarifying their values and will be used to examine participants' personal values, values attainment, and persistence towards values in the face of barriers. Part 1 asks the person to record values for 4 domains (work/education, relationships, personal growth/health, and leisure). Then, participants are asked to think of their values in each domain as "bull's eye" (the middle of the dart board). A 1 is equal to a hit in the bull's eye, which means that they are living completely in keeping with their value for that area of living. An 8 is equal to far from the bull's eye, which means that their life is way off the mark in terms of how they are living their life. Part 2 asks the person to identify obstacles to those values and rate from 1, "doesn't prevent me at all", to 7, "prevents me completely".
Time Frame: as for outcome 4
Population: SMILE Intervention arm: Work/education, relationships, personal growth/health, leisure: One participant lost to follow-up and two participants had missing data.
  SMILE Intervention arm: Obstacles: One participant lost to follow-up and four participants had missing data.
  Education Control Arm: One participant lost to follow-up, one participant died prior to completion of the A2 assessment, and one participant had missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 21 | 13
score on a scale
  Baseline: Work/Education | 4.43 (1.94) | 4.15 (1.91)
  Post-treatment: Work/Education | 4.71 (2.26) | 3.54 (1.85)
  Baseline: Leisure | 4.62 (1.88) | 3.23 (2.05)
  Post-treatment: Leisure | 4.48 (1.89) | 4.23 (1.59)
  Baseline: Relationships | 4.43 (2.29) | 3.54 (2.33)
  Post-treatment: Relationship | 4.43 (1.99) | 3.62 (2.60)
  Baseline: Personal growth/health | 4.95 (2.11) | 4.46 (2.47)
  Post-treatment: Personal growth/health | 4.95 (1.96) | 4.08 (1.98)
  Baseline: Obstacles: number analyzed (Participants) | 19 | 13
  Baseline: Obstacles | 4.89 (1.41) | 4.31 (1.80)
  Post-treatment: Obstacles: number analyzed (Participants) | 19 | 13
  Post-treatment: Obstacles | 4.32 (1.60) | 4.54 (1.51)

14. Primary Outcome: Use of Intervention Strategies
Description: Participants' use of intervention strategies will be assessed using a measure developed specific to components of the proposed intervention. Participants will be asked about how frequently treatment strategies discussed in session have been used outside of session since the previous session or last assessment depending on the timing of the questionnaire. A scale ranging from 0 "not at all" to 4 "6 or more days per week" is used.
Time Frame: Post-treatment (6-8 weeks following the baseline assessment), 4 weeks following the post-treatment/ follow-up assessment; post-treatment (6-8 weeks following the baseline assessment) reported
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE)
Number analyzed (Participants) | 20
score on a scale | 2.1 (0.97)

15. Primary Outcome: Living in Alignment With Values: The Valuing Questionnaire (VQ)
Description: The Valuing Questionnaire is a 10-item self-report questionnaire with a scale 0 = "not true at all" to 6 "completely true." Two subscale scores are calculated, Progress and Obstruction, which typically have a negative correlation. Higher scores on the Progress subscale represent a closer alignment between one's internal values and one's actions. Higher scores on the Obstruction subscale represent more interference with living consistently with one's values. The range for both subscales is 0 to 30.
Time Frame: as for outcome 4
Population: SMILE Intervention: Progress - 1 participant lost to follow-up and 2 participants with missing data at least one item of the subscale; Obstruction - 1 participant lost to follow-up and 1 participant with missing data on at least one item of the subscale
  Education Control Arm: Progress - 1 participant lost to follow-up and 1 participant died prior to completion of the A2 assessment; Obstruction - 1 participant lost to follow-up and 1 participant died prior to completion of the A2 assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm
Number analyzed (Participants) | 22 | 14
score on a scale
  Baseline: Progress: number analyzed (Participants) | 21 | 14
  Baseline: Progress | 17.05 (5.57) | 20.50 (6.04)
  Post-treatment: Progress: number analyzed (Participants) | 21 | 14
  Post-treatment: Progress | 18.43 (5.58) | 17.93 (6.66)
  Baseline: Obstruction | 13.68 (5.92) | 10.07 (6.71)
  Post-treatment: Obstruction | 9.50 (6.46) | 11.43 (6.79)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Symptom Management for Improved Physical and Emotional Wellbeing (SMILE) | Education Control Arm | Intervention Development (Patients) | Intervention Development (Caregivers) | Intervention Refinement
All-Cause Mortality (participants affected / at risk) | 1/24 | 1/16 | 1/17 | 0/13 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/16 | 0/17 | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 0/24 | 0/16 | 0/17 | 0/13 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT05593016/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT05593016/ICF_000.pdf